CLINICAL TRIAL: NCT06170827
Title: Open-Label, Single Dose, Parallel Group, Phase 1 Study in Healthy Volunteers Evaluating Safety, Tolerability, Pharmacokinetics, and Immunogenicity AIO-001 Administered by Injections
Brief Title: Study to Evaluate the AIO-001 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syneos Health (Other)
Collaborators: Aiolos Bio, Inc., a GSK Company (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-001-101
Record Dates: First submitted 2023-11-26; First posted 2023-12-14 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AIO-001 (Formulation A) (Experimental): 400 milligram (mg) of 100 milligrams per milliliter (mg/ml) AIO-001 Subcutaneous (SC) injection will be administered.
  Interventions: Drug: AIO-001
- AIO-001 (Formulation B) (Experimental): 400 mg of 182 mg/ml AIO-001 SC injection will be administered.
  Interventions: Drug: AIO-001

INTERVENTIONS:
Drug: AIO-001 — AIO-001 Solution for SC injection.

SUMMARY:
This goal of the open-label single dose study is to evaluate and compare the safety, tolerability, pharmacokinetic (PK), and immunogenicity of AIO-001 using two different formulations in 16 healthy volunteers.

DETAILED DESCRIPTION:
This is an open-label single dose, parallel group, 24-week, Phase 1 study in 16 healthy participants.

The study is designed to evaluate and compare the safety, tolerability, PK, and immunogenicity of AIO-001 using two different formulations (Formulation A and Formulation B) in 16 healthy volunteers (8 receiving each formulation).

The study will include a screening visit from Day -28 to Day -2. Eligible participants will be admitted to the clinical site on Day -1 and will be confined until completion of the assessments on Day 3. Participants will return to the clinical site for outpatient visits for study assessments and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study procedures and provide signed informed consent to participate in the study.
2. Male or female.
3. Non-smokers. Light smokers (no more than 5 cigarettes daily [approximately 50 to 60 mg of nicotine per day], or products with equivalent amount of nicotine within 3 months prior to screening) may be permitted.
4. ≥18 and ≤55 years of age.
5. BMI >18.5 and <32.0 kg/m2 and body weight ≥45.0 kg.
6. Healthy participants.

Exclusion Criteria:

1. Any clinically significant abnormal finding at physical examination at screening.
2. Clinically significant abnormal laboratory test results or positive serology test results for hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen and antibody, or QuantiFERON®-TB tuberculosis (TB) test at screening.
3. Positive pregnancy test or lactating female participant.
4. Positive urine drug screen or alcohol breath test.
5. History of anaphylaxis, or severe allergy.
6. Previous exposure to thymic stromal lymphopoietin antibody.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Nucleus Network
Locations (1):
- Q-Pharm Pty Ltd, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: Sharing Clinical Trial Data' on the GSK Study Register (www.gsk-studyregister.com).
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.

RESULTS

PARTICIPANT FLOW:
Groups:
- AIO-001: Formulation A: Participants received 400 milligrams (mg) of 100 milligrams per milliliter (mg/ml) AIO-001, administered as 4*1.0 milliliter (ml) subcutaneous (SC) injection on Day 1.
- AIO-001: Formulation B: Participants received 400 mg of 182 mg/ml AIO-001, administered as 2*1.1 ml SC injection on Day 1.
Period: Overall Study
Arm/Group | AIO-001: Formulation A | AIO-001: Formulation B
Started | 8 | 8
Completed | 7 | 7
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- AIO-001: Formulation A: Participants received 400 mg of 100 mg/ml AIO-001, administered as 4*1.0 ml SC injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | AIO-001: Formulation A | AIO-001: Formulation B | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (7.45) | 32.8 (10.48) | 33.1 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical trial participant administered a pharmaceutical product and which did not necessarily have a causal relationship with the treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. TEAEs were defined as AEs that commence on or after the time of study drug administration.
Time Frame: From Day 1 up to Day 169
Population: The safety population included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AIO-001: Formulation A | AIO-001: Formulation B
Number analyzed (Participants) | 8 | 8
Participants | 5 | 6

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital sign measurements included blood pressure, heart rate, respiratory rate, and oral temperature measurements. The clinically significant changes were based on investigator's judgement.
Time Frame: Baseline (Day -1) up to Day 169
Population: The safety population included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AIO-001: Formulation A | AIO-001: Formulation B
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in 12-lead Electrocardiogram Parameters
Description: The electrocardiogram parameters included heart rate, PR interval, QT interval, corrected QT (QTcF using Fridericia's formula) interval and QRS. The clinically significant changes were based on investigator's judgement.
Time Frame: Baseline (Day -1) up to Day 169
Population: The safety population included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AIO-001: Formulation A | AIO-001: Formulation B
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Physical Examination Findings
Description: Physical examination included assessments of the following: head, eyes, ears, nose, throat, neck, chest, lungs, abdomen, musculoskeletal, dermatological, cardiovascular/peripheral vascular, and general neurological examination. The clinically significant changes were based on investigator's judgement.
Time Frame: Baseline (Day -1) up to Day 169
Population: The safety population included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AIO-001: Formulation A | AIO-001: Formulation B
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Parameters
Description: Clinical laboratory parameters included biochemistry, hematology, and urinalysis assessment. The clinically significant changes were based on investigator's judgement.
Time Frame: Baseline (Day -1) up to Day 169
Population: The safety population included all participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AIO-001: Formulation A | AIO-001: Formulation B
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

6. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero Until the Last Observed Concentration (AUC0-last) of AIO-001
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of AIO-001. PK analysis was conducted using standard non-compartmental methods.
Time Frame: Pre-dose, 12, 24, 48, 72, 96, 120, 168, 240, 336, 504, 672, 1008, 1344, 1680, 2016, 2688, 3360, and 4056 hours post-dose
Population: The PK population included all participants who had at least 1 measured PK concentration following dosing. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*microgram per milliliter(day*mcg/mL)
Arm/Group | AIO-001: Formulation A | AIO-001: Formulation B
Number analyzed (Participants) | 7 | 7
day*microgram per milliliter(day*mcg/mL) | 4608.31 (30.04) | 4935.31 (18.18)

7. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of AIO-001
Description: Blood samples were collected at indicated time points for PK analysis of AIO-001. PK analysis was conducted using standard non-compartmental methods. The residual area was greater than 20% in 15 out of the total of 16 participants and therefore the estimation of AUC0-inf may be non-identifiable.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | AIO-001: Formulation A | AIO-001: Formulation B
Number analyzed (Participants) | 7 | 8
day*mcg/mL | 7092.12 (30.49) | 8088.05 (22.92)

8. Secondary Outcome: Maximal Observed Concentration (Cmax) of AIO-001
Description: Blood samples were collected at indicated time points for PK analysis of AIO-001. PK analysis was conducted using standard non-compartmental methods.
Time Frame: as for outcome 6
Population: The PK population included all participants who had at least 1 measured PK concentration following dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | AIO-001: Formulation A | AIO-001: Formulation B
Number analyzed (Participants) | 8 | 8
micrograms per milliliter (mcg/mL) | 43.69 (35.83) | 47.49 (22.22)

9. Secondary Outcome: Time to Maximal Observed Concentration (Tmax) of AIO-001
Description: as for outcome 8
Time Frame: as for outcome 6
Population: The PK population included all participants who had at least 1 measured PK concentration following dosing.
Measure: Median (Full Range); unit: day
Arm/Group | AIO-001: Formulation A | AIO-001: Formulation B
Number analyzed (Participants) | 8 | 8
day | 13.55 [7.94 to 21.97] | 17.43 [4.00 to 27.16]

10. Secondary Outcome: Terminal Elimination Half-life (T½) of AIO-001
Description: Blood samples were collected at indicated time points for PK analysis of AIO-001. PK analysis was conducted using standard non-compartmental methods. The residual area was greater than 20% in 15 out of the total of 16 participants and therefore the estimation of T½ may be non-identifiable.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: day
Arm/Group | AIO-001: Formulation A | AIO-001: Formulation B
Number analyzed (Participants) | 7 | 8
day | 104.34 (24.11) | 119.35 (45.20)

11. Secondary Outcome: Number of Participants With Positive Anti-drug Antibody (ADA) to AIO-001
Description: ADA-positive participant was defined as participant with at least one treatment-induced or treatment-boosted ADA-positive sample at any time during the treatment or follow-up observation period. Anti-AIO-001 antibodies were evaluated in serum samples. Serum samples were screened for antibodies binding to AIO-001.
Time Frame: Up to Day 169
Population: The immunogenicity population included all participants who received any amount of AIO-001 and had at least one post-dose ADA measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | AIO-001: Formulation A | AIO-001: Formulation B
Number analyzed (Participants) | 8 | 8
Participants | 0 | 4

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected from start of study drug administration (Day 1) up to Day 169
Description: The safety population included all participants who received at least one dose of study drug.
Arm/Group | AIO-001: Formulation A | AIO-001: Formulation B
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/8 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIO-001: Formulation A (N=8) | AIO-001: Formulation B (N=8)
COVID-19 (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Injection site pain (General disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Troponin I increased (Investigations) | 1 | 0
Myokymia (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT06170827/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT06170827/SAP_001.pdf